CLINICAL TRIAL: NCT00631995
Title: Safety and Immunogenicity of a Quadrivalent Meningococcal (A, C, Y, and W-135) Tetanus Protein Conjugate Vaccine (TetraMen-T) in Toddlers
Brief Title: Safety and Immunogenicity of a Quadrivalent Meningococcal Tetanus Protein Conjugate Vaccine in Toddlers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET32
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group 1 (Experimental)
  Interventions: Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate
- Group 2 (Experimental)
  Interventions: Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate
- Group 3 (Experimental)
  Interventions: Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate
- Group 4 (Experimental)
  Interventions: Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate
- Group 5 (Experimental)
  Interventions: Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate
- Group 6 (Active Comparator)
  Interventions: Dietary Supplement: Meningococcal polysaccharide group C conjugated

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate — 0.5 mL, Intramuscular
  Arms: Group 1
Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate — 0.5 mL, Intramuscular
  Arms: Group 2
Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate — 0.5 mL, Intramuscular
  Arms: Group 3
Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate — 0.5 mL, Intramuscular
  Arms: Group 4
Biological: Meningococcal Polysaccharide Tetanus Protein Conjugate — 0.5 mL, Intramuscular
  Arms: Group 5
Dietary Supplement: Meningococcal polysaccharide group C conjugated — 0.5 mL, Intramuscular
  Other Names: NeisVac-C® vaccine (Baxter Healthcare)
  Arms: Group 6

SUMMARY:
This study is aimed at studying quadrivalent meningococcal (A, C, Y, and W-135) Tetanus Protein Conjugate Vaccine (TetraMen-T) formulations in Toddlers.

Primary Objectives: Safety and Immunogenicity:

To describe the safety and immunogenicity profiles of:

* A single dose of each formulation of TetraMen-T vaccine
* A single dose of NeisVac-C® vaccine.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety profile and the immunogenicity response after a single dose of TetraMen-T in toddlers.

ELIGIBILITY:
Inclusion Criteria :

* Subject is healthy, as determined by medical history and physical assessment.
* Aged 12 months (± 21 days) on the day of inclusion.
* Institutional Review Board (IRB)-approved informed consent form signed by the subject's parent/legal guardian.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria :

* Serious acute or chronic disease (e.g., cardiac, renal, metabolic, rheumatologic, psychiatric, hematologic, or autoimmune disorders, diabetes, atopic conditions, congenital defects, convulsions, encephalopathy, blood dyscrasias, leukemia, lymphomas of any type, or other malignant neoplasms affecting the bone marrow or lymphatic system, acute untreated tuberculosis) that could interfere with trial conduct or completion.
* Known or suspected impairment of immunologic function.
* Acute medical illness within the last 72 hours, or temperature ≥ 37.5ºC (axillary) at the time of enrollment (temporary contraindication).
* History of documented invasive meningococcal disease or previous meningococcal vaccination.
* Known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C seropositivity as reported by the parent or legal guardian.
* Received either immune globulin or other blood products within the last 3 months, or received injected or oral corticosteroids or other immunomodulator therapy within 6 weeks of the study vaccines. Individuals on a tapering dose schedule of oral steroids lasting < 7 days and individuals (e.g., asthmatics) on a short schedule of oral steroids lasting 3 to 4 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment. Topical steroids are not included in this exclusion criterion.
* Anticipated to receive oral or injected antibiotic therapy within the 72 hours prior to the study blood draw. Topical antibiotics or antibiotic drops are not included in this exclusion criterion.
* Suspected or known hypersensitivity to any of the vaccine components.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular (IM) vaccination.
* Parent or legal guardian unable or unwilling to comply with the stu dy procedures.
* Participation in another interventional clinical trial in the 30 days preceding enrollment, or participation in another clinical trial involving the investigation of a drug, vaccine, medical procedure, or medical device during the subject's trial period.
* Diagnosed with any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the evaluation of the vaccine.
* Received any vaccine in the 30-day period prior to receipt of study vaccine, or scheduled to receive any vaccination other than influenza vaccination and hyposensitization therapy in the 30-day period after receipt of any study vaccine. Hyposensitization therapy and influenza vaccination may be received up to 14 days before or 14 days after receiving the study vaccines.
* History of seizures, including febrile seizures, or any other neurologic disorder.
* Personal or family history of Guillain-Barré Syndrome (GBS).

Ages: 12 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To provide information concerning the safety and immunogenicity after administration of TetraMenT | 30 days after each injection

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (5):
- Australia (5):
  - Herston
  - Melbourne
  - North Adelaide
  - Perth
  - Westmead

REFERENCES:
- [Result] McVernon J, Nolan T, Richmond P, Reynolds G, Nissen M, Lambert SB, Marshall H, Papa T, Rehm C. A randomized trial to assess safety and immunogenicity of alternative formulations of a quadrivalent meningococcal (A, C, Y, and W-135) tetanus protein conjugate vaccine in toddlers. Pediatr Infect Dis J. 2012 Jan;31(1):e15-23. doi: 10.1097/INF.0b013e31823e1e34. PMID 22094636
- See also: Related Info — http://www.sanofipasteur.com